CLINICAL TRIAL: NCT02434965
Title: A Safety and Feasibility Study of Autologous Cord Blood (CB) and Human Placental Derived Stem Cells (HPDSC) in Neonates With Severe Hypoxic-Ischemic Encephalopathy (HIE)
Brief Title: Autologous Cord Blood and Human Placental Derived Stem Cells in Neonates With Severe Hypoxic-Ischemic Encephalopathy
Acronym: HPDSC+HIE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not started
Sponsor: New York Medical College (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-554
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2019-09

CONDITIONS: Severe Hypoxic-ischemic Encephalopathy
Keywords: Neonates; hypoxic-ischemic encephalopathy; human placental-derived stem cells; autologous
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Cord Blood and HPDSC (Experimental): Autologous cord blood and placental blood will be collected after birth of child and administered in divided aliquots during the first week of life.
  Interventions: Drug: HPDSC; Drug: Cord blood

INTERVENTIONS:
Drug: HPDSC — Autologous HPDSC collected after birth will be infused in aliquots. one-half of the HPDSC infused on Day 2; one-half of the collected HPDSC will be infused on Day 8.
Drug: Cord blood — Autologous Cord Blood collected after birth will be infused in aliquots. One-third of the collected cord blood will be infused within the first 24 hours after birth (Day 0); one-third of the collected cord blood will be infused on day 3; and one-third of the collected cord blood unit will be infused on Day 7.

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of autologous human placental-derived stem cells (HPDSC) in combination with autologous cord blood in neonates with severe hypoxic-ischemic encephalopathy.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the safety, tolerability and feasibility of intravenous administration of autologous cord blood (CB) and autologous human placental derived stem cells (HPDSC) in neonates with severe hypoxic-ischemic encephalopathy (HIE). It is hypothesized that the administration of autologous CB and autologous HPDSC will be safe and well tolerated in neonates with severe HIE.

Additionally, postnatal neuro-developmental outcomes in neonates with HIE after autologous CB and HPDSC therapy will be measured; HIE injury to the neonate/infant brain post autologous CB and HPDSC therapy by imaging will be characterized; the pluripotent stem cell properties of CB and HPDSC will be characterized; serum levels of selected circulating cytokine and neurotrophic factors in neonates with HIE before and after autologous CB and HPDSC therapy will be compared and immune cell phenotype and function in neonates with HIE before and after autologous CB and HPDSC therapy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 36 weeks
* Birth weight ≥ 1800 grams
* Postnatal age after birth of less than 6 hours
* Autologous cord blood and HPDSCs available for infusion
* Plus one or more of the following criteria: Apgar ≤ 5 at 10 minutes of postnatal age, or Continued need for resuscitation ≥10 min after birth, or Acidosis-cord blood pH or arterial blood pH within 60 minutes of birth ≤ 7.0 pH, or Base deficit ≥ minus 16mEq in cord blood and within 60 min of birth.
* Plus Moderate to Severe Altered State of Consciousness, by one or more of the following: Hypotonia, or Abnormal reflexes, or Absent/weak suck.

Exclusion Criteria:

* Major life-threatening or surgical anomalies
* Polycythemia (hematocrit > 65%)
* Congenital infection based on antenatal diagnosis of TORCH infection
* Parental refusal for study
* Infant expected to live < 24h, medical care is considered futile and no additional therapy will be offered by the attending neonatologist

Ages: 1 Minute to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with infusion reaction as a measure of safety and tolerability | within the first 30 days
  Any infusion reaction to autologous human placental-derived stem cells (HPDSC) administered in conjunction autologous cord blood in neonates with severe hypoxic-ischemic encephalopathy will be assessed for safety and tolerability

SECONDARY OUTCOMES:
Improvement in neurological condition | 2 years post HPDSC infusion
  Improvement in neurological condition as shown on head MRI, DTI and neurological development by Sarnat testing.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No
Study not enrolling